CLINICAL TRIAL: NCT04189900
Title: Generation of Biological Samples Positive to Triptorelin for Anti-doping Control
Acronym: TRIPTO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IMIMFTCL/TRIPTO
Record Dates: First submitted 2019-12-04; First posted 2019-12-06 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Healthy Volunteers
Keywords: Triptorelin; Anti-doping control; Athletic performance; Gonadotropin-releasing hormone
MeSH Terms: interventions — Triptorelin Pamoate

STUDY DESIGN:
Intervention Model Description: The study model consists on a single group of subjects who receive the treatment condition (triptorelin)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Triptorelin (Experimental): The subjects in this group receive a single dose treatment. Biologic sample collection (urine) from 48 hours pre-administration to 48 hours post administration.
  Interventions: Drug: Triptorelin

INTERVENTIONS:
Drug: Triptorelin — Subjects receive a single subcutaneous dose of 0,1 mg of Triptorelin acetate.

SUMMARY:
Background:

Androgens are used for doping purpose because they can increase muscle mass and strength. These drugs are included in the list of prohibited substances of the World Anti-Doping Agency (WADA). The prohibition of its use has given rise to a great variety of strategies of indirect androgenic doping, whose purpose is to produce a sustained increase in endogenous testosterone.

Triptorelin acetate is a gonadotropin-releasing hormone (GnRH) agonist. Daily subcutaneous administration of triptorelin causes an initial increase in circulating levels of luteinizing hormone (LH) and follicle stimulating hormone (FSH), producing a transient increase in testosterone levels. However, prolonged daily administration results in a paradoxical decrease in LH and FSH levels due to desensitization of GnRH receptors, decreasing testosterone production to levels similar to castration.

Thus, the initial flare reaction produced by triptorelin administration could be used by athletes as an indirect androgenic doping method to stimulate the synthesis of endogenous LH and testosterone with the aim of improving physical performance.

Hypothesis:

Subcutaneous administration of triptorelin in healthy subjects allows obtaining positive urine samples that will be used to identify analytical strategies for doping detection. Triptorelin concentrations and its metabolites can be measured in urine.

Objectives:

Primary objective: To measure triptorelin concentrations in urine samples for anti-doping control.

Secondary objectives: To identify triptorelin metabolites in urine. To explore the time window in which the drug or its metabolites can be detected in urine after administration.

Methods:

Phase I, open, non-randomized, uncontrolled clinical trial, with a treatment condition (triptorelin) administered subcutaneously in a single dose to 2 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male volunteers aged between 18 and 45 years.
* Able to understand and accept the trial procedures and able to sign an informed consent.
* History and physical examination that demonstrate not presenting organic or psychiatric disorders.
* ECG, blood and urine tests performed at screening should be within normal limits. Minor or punctual variations of these limits of normality are admitted if, in the opinion of the Principal Investigator, they have no clinical significance, do not pose a risk to the subject and do not interfere with the evaluation of the product. These variations and their non-relevance will be justified in writing specifically.
* Body mass index (weight/size^2) between 19 and 25 kg/m2, and weight between 50 and 90 kg. BMI between 25 and 27 kg/m2 may be included at the discretion of the Principal Investigator.

Exclusion Criteria:

* Failure to meet the inclusion criteria.
* History of allergy, idiosyncrasy, hypersensitivity or adverse reactions to the active substance or similar nonapeptides and to any of the excipients.
* Serious adverse reactions to other medications.
* Subjects with contraindications to treatment with the study drug (according to Summary of Product Characteristics).
* Background or clinical evidence of psychiatric disorders, alcoholism, drug abuse or addiction to other substances (except for nicotine) or regular consumption of psychoactive drugs.
* Having participated in another clinical trial with medication in the three months prior to the start of the study.
* Having donated blood during the two months prior to the start of the study.
* Having suffered an organic disease or major surgery in the six months prior to the start of the study.
* Background or clinical evidence of cardiovascular, respiratory, renal, hepatic, endocrine, gastrointestinal, hematological, neurological or other acute or chronic diseases that, in the opinion of the Principal Investigator or the collaborators designated by him, may pose a risk to the subjects or interfere with the objectives of the study. Especially epileptic seizures or history of epilepsy.
* Have taken medication regularly in the month prior to the study sessions, with the exception of vitamins, herbal remedies or dietary supplements that, in the opinion of the Principal Investigator or the collaborators designated by him, do not pose a risk to the subjects and do not interfere with the objectives of the study. Treatment with single doses of symptomatic medication in the week prior to the study session will not be exclusive if it is assumed that it has been completely eliminated on the day of the experimental session.
* Smokers of more than 20 cigarettes daily the 3 months prior to the study.
* Consumption of more than 40 g of alcohol daily.
* Consumers of more than 5 coffees, teas, cola drinks and/or other stimulant drinks (xanthines) per day in the 3 months prior to the start of the study.
* Being unable to understand the nature of the trial and the procedures requested to follow.
* Positive serology for hepatitis B, C or HIV.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Urine concentration of triptorelin | 0-4 hours post-administration
  Concentration of triptorelin in urine sample (Fraction 1)
Urine concentration of triptorelin | 4-8 hours post-administration
  Concentration of triptorelin in urine sample (Fraction 2)
Urine concentration of triptorelin | 8-12 hours post-administration
  Concentration of triptorelin in urine sample (Fraction 3)
Urine concentration of triptorelin | 12-24 hours post-administration
  Concentration of triptorelin in urine sample (Fraction 4)
Urine concentration of triptorelin | 24-48 hours post-administration
  Concentration of triptorelin in urine sample (Fraction 5)

SECONDARY OUTCOMES:
Urine concentration of triptorelin metabolites | 0-4 hours post-administration
  Concentration of triptorelin metabolites in urine sample (Fraction 1)
Urine concentration of triptorelin metabolites | 4-8 hours post-administration
  Concentration of triptorelin metabolites in urine sample (Fraction 2)
Urine concentration of triptorelin metabolites | 8-12 hours post-administration
  Concentration of triptorelin metabolites in urine sample (Fraction 3)
Urine concentration of triptorelin metabolites | 12-24 hours post-administration
  Concentration of triptorelin metabolites in urine sample (Fraction 4)
Urine concentration of triptorelin metabolites | 24-48 hours post-administration
  Concentration of triptorelin metabolites in urine sample (Fraction 5)

CONTACTS AND LOCATIONS:
Overall Officials: Ana M Aldea Perona, Dr, Study Director — IMIM (Hospital del Mar Medical Research Institute)
Locations (1):
- IMIM (Hospital del Mar Medical Research Institute), Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No